CLINICAL TRIAL: NCT01910948
Title: Efficacy of Perioperative Application of Omega-3 Polyunsaturated Fatty Acids on Postoperative Immunization in Gastric Cancer Patients - A Prospective, Randomized Clinical Trial
Brief Title: Perioperative Application of Omega-3 Polyunsaturated Fatty Acids in Gastric Cancer Patients
Acronym: PAOPUFAGC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jian Suo (Other)
Responsible Party: Sponsor-Investigator, Jian Suo, Headmaster, Dept.of General Surgery, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: omega-3 PUFA
Record Dates: First submitted 2013-07-23; First posted 2013-07-30 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Gastric Cancer
Keywords: omega-3 gastric cancer perioperation
MeSH Terms: conditions — Stomach Neoplasms | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- omega-3 polyunsaturated fatty acids (Experimental): The included patients will be randomly divided into two groups A and B, two groups of patients 4 days before operation begin to give parenteral nutrition: A: the control group of normal intravenous nutrition. B: the trial group,add omega-3 polyunsaturated fatty acids 0.2 g/kg to parenteral nutrition, no use on the day of surgery, postoperative 2 days continue to add omega-3 polyunsaturated fatty acids 0.2 g/kg.
  Interventions: Drug: omega-3 polyunsaturated fatty acids

INTERVENTIONS:
Drug: omega-3 polyunsaturated fatty acids — The included patients will be randomly divided into two groups A and B, two groups of patients 4 days before operation begin to give parenteral nutrition: A: the control group of normal intravenous nutrition. B: the trial group,add omega-3 polyunsaturated fatty acids 0.2 g/kg to parenteral nutrition, no use on the day of surgery, postoperative 2 days continue to add omega-3 polyunsaturated fatty acids 0.2 g/kg.
  Other Names: omega-3 PUFA; ω-3 PUFA

SUMMARY:
To evaluate immunomodulatory effects of perioperative application of omega-3 polyunsaturated fatty acids in gastric cancer surgery, the effects of postoperative recovery, the improvement of nutritional status, incidence rate of related complications, and whether it can reduce the average postoperative hospitalization days.

DETAILED DESCRIPTION:
Methods: Choose from 6 to 2013-2013-12 gastric cancer patients, according to inclusion criteriaS to choose the objectS of study from the gastric cancer patients coming to our hospital 2013-06 to 2013-12 .The included patients will be randomly divided into two groups A and B, two groups of patients 4 days before operation begin to give parenteral nutrition: A: the control group of normal intravenous nutrition. B: the trial group,add Omega-3 Polyunsaturated Fatty Acids 0.2 g/kg to parenteral nutrition, no use on the day of surgery, postoperative 2 days continue to add Omega-3 Polyunsaturated Fatty Acids 0.2 g/kg. Detect and compare CRP、TNF-α、IL-1、IL-4、lL-6、 IL-8、lL-10 levels of two groups in days before parenteral nutrition and applicating 3rd day and postoperative 1st, 3rd, 5th,and detect liver function in preoperative and postoperative 2nd,5th,7th day. Record postoperative anal exhaust time, postoperative complications, postoperative hospital days, preoperative and postoperative body weight.Results: Trail group patients compared with the control group,Omega-3 Polyunsaturated Fatty Acids can reduce early postoperative inflammatory cytokines release, reduce the postoperative fever time, reduce the incidence of systemic inflammatory response syndrome, promote the recovery of gastrointestinal function, improve the nutritional state of patients, reduce infection and related complications after the surgery and reduce postoperative hospitalization days. Conclusions: Perioperative application of omega 3 PUFA can reduce the release of inflammatory cytokines, regulating cell and humoral immunity, reduce the postoperative fever time, reduce the local inflammation medium that inhibit the gastrointestinal peristalsis, promote the recovery of gastrointestinal function, improve the nutritional state of patients, thereby reducing the occurrence of postoperative infection and related complications, reduce postoperative hospitalization days.

ELIGIBILITY:
Inclusion Criteria:

* Patients coming to FirstJilinU diagnosed gastric cancer by endoscopy and pathology.
* No preoperative treatment, the gastric cancer radical surgery in our hospital is the first treatment.
* Nutrition screening score (NRS 3 or higher).
* Albumin and (or) immune enhancer were not used within two weeks before operation .
* No blood system diseases.

Exclusion Criteria:

* Being in the acute phase of inflammation before operation and emergency surgery.
* Patients combined metabolic diseases such as diabetes, hyperthyroidism, immune system disease or taking immunosuppressants;
* Combined hepatic insufficiency.
* Spleen resected in operation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-06; Primary Completion 2013-12 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
blood immune factors | 10 days